CLINICAL TRIAL: NCT00816335
Title: Pilot Study Evaluating a Combined and Integrated Technological Approach of F-18-FDG-Directed Perioperative PET/CT Imaging and Intraoperative Handheld Gamma Prove Detection of Known and Occult Disease in Patients Undergoing Surgery for Solid Malignancies
Brief Title: Fludeoxyglucose F 18 PET/CT Imaging in Finding Cancer in Patients Undergoing Surgery for Solid Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Stephen Povoski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-08031; NCI-2012-00958 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): F-FDG-directed surgery for known or suspected malignancy using gamma detection probes.
  Interventions: Procedure: PET/CT scan; Drug: 18F-FDG Injection; Procedure: Preoperative 18F-FDG PET/CT Scan; Drug: 18F-FDG for patients with Bladder Cancer; Procedure: Surgical Procedure; Procedure: Specimen PET/CT Scan

INTERVENTIONS:
Procedure: PET/CT scan — For all patients undergoing a preoperative PET/CT scan on the day of surgery, at approximately 70 minutes post-injection of 18F-FDG, a diagnostic whole body PET/CT scan will be obtained on a Siemens Biograph 16 PET/CT scanner (Siemens, Knoxville, TN).
  Other Names: Positron emission tomography; Computed tomography
Drug: 18F-FDG Injection — Patients undergoing a preoperative PET/CT scan the day of surgery, are required to have fasted for at least 4 hours prior to the anticipated preoperative PET/CT scan. Patients participating in this pilot study (whether they have had their preoperative PET/CT scan prior to the day of surgery or whether they are having their preoperative PET/CT scan on the day of surgery) will receive a preoperative IV injection into a peripheral vein of 15 mCi of 18FFDG at time interval of approximately 60 to 180 minutes prior to anticipated time of surgery.
  Other Names: Fludeoxyglucose; fdg
Procedure: Preoperative 18F-FDG PET/CT Scan — Patients undergoing preoperative PET/CT scan day of surgery, at approximately 70 minutes post-injection of 18F-FDG, a diagnostic whole body PET/CT scan will be obtained. PET imaging will immediately be preceded by noncontrast transmission CT (for attenuation correction and anatomic correlation purposes) and will be obtained from the base of the skull to the mid thighs. Bed positions will be scanned for 3 minutes each, moving the patient through the scanner in a craniocaudal direction. Once the preoperative PET/CT scan is acquired, images will be reviewed by the nuclear medicine physician and the surgeon.
  Other Names: Fludeoxyglucose; fdg; Positron emission tomography; Computed tomography
Drug: 18F-FDG for patients with Bladder Cancer — Elimination of 18F-FDG by the urinary system and accumulation in the bladder impacts the differentiation between residual 18F-FDG in the bladder and activity in tumor and adjacent lymph nodes. For patients with bladder cancer, the urinary catheter routinely placed in the operating room will be inserted in the Ambulatory Surgery Unit (ASU) by the urologist on-service or the urology research nurse. A 3-way Foley catheter will be placed for continuous bladder irrigation with Normal Saline (0.9%) initiated in ASU and will continue for the duration of the imaging procedure at a standard rate of 10cc/minute. The urology research nurse will transport the patient to and from the PET/CT area and monitor the continuous bladder irrigation during the imaging session.
  Other Names: Fludeoxyglucose; fdg
Procedure: Surgical Procedure — Previously determined operative procedure based on type of solid malignancy. Factors include extent and location of disease, physiologic status of patient intraoperatively, any technical considerations influenced by anatomic constraints, and a risk: benefit analysis of proposed procedure. The decision to proceed with resection on these factors, and will constantly re-evaluate during resection to ensure patient well-being, both short and long term, is foremost consideration. Evaluation of extent of disease during surgical exploration will include inspection and palpation of entire area being evaluated. Tissue that is highly suspicious for involvement with metastatic disease that alters the surgical decision making plan of resection will be biopsied or resected for histologic confirmation if feasible and safe. If patient is found to have resectable disease, deemed safe patient, surgeon will continue and proceed with definitive surgical resection with assistance of handheld gamma probe.
Procedure: Specimen PET/CT Scan — Resected surgical specimen will be placed on top of paraffin block. Digital photos of the specimen will be obtained for visual correlation of specimen placement on paraffin block. Two bed position 10 minute specimen PET/CT scan will be performed on surgical specimen. If remnant tissue is available, a second image maybe acquired via MRI. Images will be processed and reviewed for quality and presence or absence of hypermetabolic foci and correlated with anatomical information provided by CT and MRI imaging that were originally noted in the preoperative clinical PET/CT scan. During the time when the excised surgical specimens are transported to radiology for specimen PET/CT scanning, additional evaluation of these ex-vivo specimens with other tumor detection devices may be undertaken. Specimen will then be transported back to the operating room in order to be sent to and processed by surgical pathology for standard pathologic evaluation.

SUMMARY:
The purpose of this pilot study is to evaluate a combined and integrated technological approach of 18F-FDG-directed perioperative PET/CT imaging and intraoperative handheld gamma probe detection of known and occult disease in patients undergoing surgery for solid malignancies.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To determine if the perioperative PET/CT imaging (consisting of preoperative PET/CT imaging, specimen PET/CT imaging, and postoperative PET/CT imaging) combined with intraoperative use of the handheld gamma probe is feasible during a surgical procedure to resect malignancy.
2. To evaluate if perioperative PET/CT imaging can assist in intraoperatively localizing tumor and verify complete resection of disease.
3. To evaluate intraoperative detection of tumor sites using a handheld gamma probe after preoperative injection of 18F-FDG combined with preoperative PET/CT imaging.
4. To evaluate specimen PET/CT imaging using the preoperative 18F-FDG dose for detecting presence of tumor within the specimen and for assessing surgical margins.
5. To evaluate specimen MRI imaging for detecting presence of tumor within remnant tissue of appropriately selected resected specimens and for assessing surgical margins.
6. To evaluate standard pathology sampling with image guided pathology sampling (using specimen PET/CT imaging) in order to determine if sensitivity and accuracy of pathologic evaluation may be improved with PET/CT image guidance.
7. To compare activity of surgical specimen samples in a well counter and correlate activity with pathologic findings and tumor burden in order to determine if the concepts in the previous two specific aims can be utilized to benefit patients treated at centers without access to PET/CT imaging equipment.

OUTLINE: Patients undergo pre- and postoperative fludeoxyglucose F 18 (^18FDG) PET/CT imaging. An intraoperative handheld gamma probe is used to detect ^18FDG-avid tissues. Resected specimens are assessed by ^18FDG PET imaging for intraoperative verification of complete tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.
* Patients must either have a histologic-confirmed solid malignancy or have a suspected solid malignancy which has required a diagnostic preoperative PET/CT scan or for which a diagnostic preoperative PET/CT scan has been recommended
* Patients must clinically have been determined to be a candidate for the indicated surgical procedure.
* Patients may have had prior surgery and/or chemotherapy with no limit to the number of prior therapeutic procedures or chemotherapeutic regimens.
* Patients must have a performance status of 0, 1 or 2 by ECOG standards.
* Patients must give written informed consent, including consent to have IV line placed for 18F-FDG administration.
* Females of childbearing age must have a negative pregnancy test (by Beta HCG qualitative analysis), must have had a history of a surgical sterilization, or must give history of no menses in past twelve months.
* Fasting blood sugar less than 200 mg/dl.

Exclusion Criteria:

* Any patient with active CNS tumor involvement.
* Any patient who is pregnant or lactating.
* Any patient with a body size and habitus that is determined to prohibit use of the diagnostic equipment.
* Any patient with a tumor burden that is determined to be so great (as determined by preoperative PET/CT scanning or intraoperative findings) that further surgery is not advised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Determine perioperative PET/CT imaging combined with intraoperative use of handheld gamma probe is feasible during surgical procedure to resect malignancy. | up to five years

SECONDARY OUTCOMES:
Evaluate if perioperative PET/CT imaging can assist in intraoperatively localizing tumor and verify resection of disease. | up to five years
Evaluate intraoperative detection of tumor sites using a handheld gamma probe after preoperative injection of 18F-FDG combined with preoperative PET/CT imaging. | up to five years
Evaluate specimen PET/CT imaging using the preoperative 18F-FDG dose for detecting presence of tumor within the specimen and for assessing surgical margins. | up to five years
Evaluate specimen MRI imaging for detecting presence of tumor within remnant tissue of appropriately selected resected specimens and for assessing surgical margins. | up to five years
Evaluate standard pathology sampling with image guided pathology sampling (using specimen PET/CT imaging) in order to determine if sensitivity and accuracy of pathologic evaluation may be improved with PET/CT image guidance. | up to five years
Compare activity of surgical specimen samples with pathologic findings and tumor burden in order to determine if the concepts in previous two specific aims can be utilized to benefit patients treated at centers without access to PET/CT imaging equipment. | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Povoski, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Povoski SP, Chapman GJ, Murrey DA Jr, Lee R, Martin EW Jr, Hall NC. Intraoperative detection of (1)(8)F-FDG-avid tissue sites using the increased probe counting efficiency of the K-alpha probe design and variance-based statistical analysis with the three-sigma criteria. BMC Cancer. 2013 Mar 4;13:98. doi: 10.1186/1471-2407-13-98. PMID 23496877
- See also: Jamesline — http://cancer.osu.edu